CLINICAL TRIAL: NCT07016152
Title: An Open-label, Dose-finding, Phase I Study to Evaluate the Safety and Immunogenicity of a Bivalent Klebsiella Pneumoniae Vaccine (CHO-V08) in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cho Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: KLEBBI-001
Record Dates: First submitted 2025-06-02; First posted 2025-06-11 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Klebsiella Pneumoniae Infection; Vaccine
Keywords: Klebsiella Pneumoniae Infection; Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- low dose (CHO-V08) (Experimental)
  Interventions: Biological: Glyconjugate Klebsiella pneumoniae bivalent vaccine
- high dose (CHO-V08) (Experimental)
  Interventions: Biological: Glyconjugate Klebsiella pneumoniae bivalent vaccine

INTERVENTIONS:
Biological: Glyconjugate Klebsiella pneumoniae bivalent vaccine — CHO-V08 is a glycoconjugate bivalent vaccine in sterile suspension.

SUMMARY:
CHO-V08 is currently being developed as a prevention vaccine against nosocomial and community-acquired infection caused by hypervirulent Klebsiella pneumoniae K1 and K2 serotypes. The goal of study (KLEBBI-001) is to evaluate the safety, reactogenicity, and immunogenicity of the preventive vaccine of CHO-V08 in healthy volunteers aged from 18 to 50 years old.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female, aged 18 to 50 years old (inclusive) for Cohorts 1 and 2 at the Screening visit.
* Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive) at the Screening visit.
* Physically and mentally capable of participating in the study and willing to adhere to study procedures.
* Able to provide signed informed consent.
* In generally good health by medical history, physical examination, vital signs, and clinical laboratory findings at the Screening visit based on the investigator's judgment.
* Negative serology test for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, and hepatitis C antibody at the Screening visit.
* Female subject with childbearing potential must have a negative result of pregnancy test at the Screening visit.
* Female subject with childbearing potential must be willing to implement adequate, highly effective contraceptive measure during the study period.
* Male subject who agrees to use an adequate method of contraception during the study period.

Exclusion Criteria:

* Any medical or psychiatric condition that, in the opinion of the investigator, may interfere with optimal participation in the study or place the subject at increased risk of AEs.
* Suspected or known hypersensitivity (including allergy) to any of the vaccine components.
* History of hypersensitivity or allergy to any vaccine, especially pneumococcal vaccine.
* Current or previous, confirmed, or suspected disease caused by Klebsiella pneumoniae.
* Medical conditions as a contraindication to the intramuscular vaccination and blood draws, e.g., coagulation disorder.
* Any abnormality or permanent body art (e.g., tattoo) that would interfere with the observation of local reactions at the injection site (deltoid region).
* Acute or chronic, clinically significant cardiovascular, pulmonary, hepatic or renal diseases and/or insufficiency as determined by physical examination or laboratory tests.
* Known or suspected impairment of immunological function, e.g., asplenia/splenectomy or history of autoimmune/immune-mediated diseases or lymphoproliferative disorders.
* Any screening laboratory abnormalities that are Grade 2 or above or deemed clinically significant in the opinion of the investigator.
* Subjects with an electrocardiogram (ECG) at the Screening visit that demonstrates clinically relevant abnormalities which may affect subject safety or study results in the opinion of the investigator.
* Positive test for SARS-CoV-2 virus at the Screening visit.
* Use of any antibiotic therapy within 1 week prior to the first study vaccination.
* History of any chronic or progressive disease that, according to judgment of the investigator, could interfere with the study outcomes or pose a threat to the subject's health.
* History of cancer (except localized skin cancer without metastases) within 5 years prior to the Screening visit.
* History or presence of heavy smoking (defined as > 10 cigarettes per day; approximately half pack per day) as documented in medical chart or by verbal confirmation at the Screening visit.
* Documented history of substance or alcohol abuse in the medical chart or by verbal confirmation within 6 months prior to the Screening visit.
* Received any vaccination (live, inactivated, or bacterial) within 1 month prior to the Screening visit and plans to receive vaccination within 4 weeks after the last study vaccination during the study period. Exception can be made with marketed vaccines against seasonal influenza or COVID-19 outside the 28-day window of the study vaccination.
* Received major surgery or radiation therapy within 3 months prior to the Screening visit.
* Onset of influenza-like illness as defined by: fever (temperature ≥ 38℃), dry cough, headache, fatigue, respiratory sputum production, dysgeusia, anosmia, shortness of breath, muscle and joint pain, or sore throat within 1 week prior to the Screening visit.
* Female subject who is pregnant or lactating at the Screening visit or plans to be pregnant during the study period or lactate from the time of the first vaccination through 60 days after the last vaccination.
* Received any investigational drug or device or have participated in a clinical study within 3 months prior to the Screening visit.
* Any confirmed or suspected abnormal immune function, immunosuppression, or immunodeficiency or received any immunosuppressants (including systemic corticosteroids) or immunomodulators within 3 months prior to the Screening visit.
* Had blood donation within 2 weeks prior to the Screening visit.
* Received any blood products or immunoglobulin within 3 months prior to the Screening visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-11-05 (Estimated); Study Completion 2027-04-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and reactogenicity of the CHO-V08 vaccination. | 1 year
  Occurrence, severity, and relationship of immediate adverse reactions, solicited, unsolicited adverse events following each vaccination. Occurrence, severity, and relationship of medically-attended AEs (MAAEs), adverse events of special interest (AESIs), new-onset chronic medical conditions (NOCMCs), and serious adverse events (SAEs) through the study completion.

SECONDARY OUTCOMES:
To assess the immunogenicity of immunoglobulins M and G (IgM and IgG) following the CHO-V08 vaccination. | 1 year
  1. Geometric mean titer (GMT) of Kp serotype specific IgM and IgG antibody titers.
  2. Seroconversion rate (SCR) in Kp serotype specific IgG antibody titers from baseline.
  3. The geometric mean fold rise (GMFR) in Kp serotype specific IgM and IgG antibody titers from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital- Clinical Trial Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No